CLINICAL TRIAL: NCT06242626
Title: Low T3 Versus Low T3T4 Syndrome in Septic Shock Patients- a Prospective Observational Cohort Study
Brief Title: Euthyroid Sick Syndrome in Septic Shock
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital Zenica (Other)
Responsible Party: Principal Investigator, Mirza Kovacevic, Principal Investigator, Cantonal Hospital Zenica
Other Study IDs: ESS2
Record Dates: First submitted 2023-12-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low T3
  Interventions: Other: observation
- Low T3T4
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — analysis of clinical, laboratory and haemodynamics parameters

SUMMARY:
This prospective observational cohort study included all septic shock patients with two groups of ESS and anylised in 28-day outcome, clinical biochemical parameters and hemodynamic monitoring.

DETAILED DESCRIPTION:
This prospective observational cohort study was conducted between October 2022 and August 2023 after the institutional ethics committee's approval (N0 00-03-35-38-14/22) and patients' written consent, registered at ClinTrials.gov (NCT). Inclusion criteria were all septic shock patients with ESS with absence of previous pituitary and thyroid disease. Exclusion criteria were: age below 18, patients with previous thyroid disease or an enlarged thyroid gland, pregnant women and patients who refused to participate in the study.

Patients and study protocol Upon admission to the ICU, patients who met the criteria for septic shock according to Surviving Sepsis Campaign and the criteria for ESS were divided into two groups: group 1 - low T3 and group 2 - low T3T4.

Definitions Septic shock is defined as a consequence of sepsis, characterized by hypotension requiring the use of vasopressors to achieve mean arterial pressure (MAP) ≥65 mmHg after crystalloid resuscitation and lactate values >2 mmol/L [14].

ESS is an abnormal finding of thyroid hormones in the absence of a previous disorder of hypothalamic-pituitary and thyroid function. The most common changes are low T3, followed by low T3 and T4 with normal TSH [15]. All patients included in the study were treated according to the Sepsis Survival Campaign guidelines from 2016 [16].

Data collection Demographic data with mortality scores (APACHE II (Acute Physiology And Chronic Health Evaluation II), SAPS II (Simplified Acute Physiology Score II) and SOFA (Sequential Organ Failure Assessment) score were collected on the admission in the ICU.

Laboratory parameters were analysed on the day of admission (T0), on the first (T1) and third (T2) day of ICU stay, and included analysis of complete blood count, C-reactive protein (CRP), procalcitonin (PCT), differential blood count, acid-base status with lactates, albumins and thyroid hormones: TSH (thyroid-stimulating hormone), FT3 (free triiodothyronine), FT4 (free thyroxine). Hemodynamic monitoring included monitoring of arterial blood pressure (systolic pressure (SBP), mean pressure (MAP), diastolic pressure (DBP)) and heart rate every hour during the first 4 days. Vasoactive drug requirement were expressed through the vasoactive drug-dependent index (VDI) and the shock index (SI), and calculated as follows:

VDI: ((dobutamine dose × 1) + (norepinephrine dose × 100) + (vasopressin dose × 100) + (epinephrine dose × 100))/MAP SI: heart rate/systolic blood pressure Mechanical ventilation requirement is categorized as YES or NO, the length of ICU stay is expressed in days and 28-day survival and characterized as transfer or death.

ELIGIBILITY:
Inclusion Criteria:

* septic shock patients,
* euthyroid sick syndrome

Exclusion Criteria:

* age below 18,
* patients with previous thyroid disease or an enlarged thyroid gland,
* psychiatric patients,
* pregnant women or women who gave birth in the past 6 months and
* patients who refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty seven patients who met criteria for septic shock according to new definitions according to Surviving Sepsis Campaign and criteria for euthyroid sick syndrome were divided into two groups: group 1 - low T3 and group 2 - low T3T4
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  28-day outcome noted as discharge from the ICU or death
blood pressure | 4 days
  Monitoring of arterial blood pressure (systolic pressure (SBP), mean pressure (MAP), diastolic pressure (DBP)) during the first 4 days in the ICU expressed in mmHg
heart rate | 4 days
  Monitoring of heart rate during the first 4 days in the ICU expressed in beats/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Mirza Kovacevic, Zenica, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No